CLINICAL TRIAL: NCT00135044
Title: A Randomised Double Blind Controlled Crossover Trial of Intravenous Taurine Supplementation in Parenteral Nutrition as an Effective Treatment for Reducing Hepatobiliary Complications in Chronic Intestinal Failure
Brief Title: A Trial of Taurine Supplementation in Parenteral Nutrition 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Fresenius AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Taurine05
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Cholestasis
Keywords: taurine; intestinal failure; HPN; hepatobiliary complications; chronic intestinal failure (CIF)
MeSH Terms: conditions — Cholestasis; Intestinal Failure | interventions — Dietary Supplements

INTERVENTIONS:
Procedure: intravenous taurine in nutritional supplement

SUMMARY:
The purpose of this study is to investigate whether the inclusion of 1g of intravenous taurine as part of the nitrogen source of parenteral nutrition reduces parenteral nutrition associated cholestatic liver disease, a common side effect of parenteral nutrition.

DETAILED DESCRIPTION:
Parenteral nutrition associated cholestasis (PNAC) is one of the main causes of death during long-term home parenteral nutrition (HPN). In one study 65% of patients on NPN developed PNAC after a median of 6 months and 41.5% developed HPN associated liver disease after a median of 17 months. It is thought that this condition develops due to changes in bile acid conjugation. Bile acids are conjugated with either taurine or glycine before their secretion in bile. Man obtains taurine mostly from the diet and hepatic taurine conjugation of bile acids accounts for 30-40% of the total bile acid pool. Taurine-conjugated bile acids are more water soluble and less toxic than glycine-conjugated bile acids. The ratio of glycine to taurine conjugated bile acids appears to be important and studies in rats have found that the bile acid sulfolithocholate, which is conjugated with glycine, was cholestatic while the taurine conjugated was not. Further studies in guinea pigs have shown that dietary taurine supplements prevent the cholestasis induced by sulfolithocholate by increasing the percentage of taurine conjugated bile acids. Patients on intravenous nutrition with intestinal failure may not re-absorb bile acids normally and may have increased losses of taurine conjugated of bile acids. They have also been found to have low levels of taurine. It is thought that chronic taurine deficiency, by altering the pattern of conjugation of bile acids, may predispose to cholestasis and ultimately severe hepatic dysfunction. In a study of hepatobiliary surgical patients given dietary taurine post operatively, there was enhanced conjugation and secretion of bile acids. Bilirubin levels fell during taurine supplementation compared to patients not receiving taurine although this was not significant. We are going to investigate if parenteral taurine supplementation is beneficial in our patients experiencing this condition.

ELIGIBILITY:
Inclusion Criteria:

* Chronic intestinal failure (CIF) patients on long term home parenteral nutrition, under the care of the Nutrition and Intestinal Failure Clinic at St Mark's, who have PNAC.
* Must be over 18
* On HPN for 6 months and stable
* Life expectancy of over 12 months
* HPN should provide > 75-80% of estimated nutritional requirements
* Should be on HPN for 5 or more days per week

Exclusion Criteria:

* No consent.
* Pregnancy/lactation.
* Planned surgery.
* Renal failure.
* Hepatitic failure, ultrasound proven fibrosis or cirrhosis, poorly controlled diabetes, hepatitis B or C, autoimmune liver disease, receiving > 40 kcal/kg/day from HPN, current sepsis, co-existing surgical complications such as intestinal obstruction, hepatotoxic drugs, primary liver cancer or metastases or any other cause for pre and post hepatic jaundice.

Inability to adhere to the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-06

PRIMARY OUTCOMES:
Whether the inclusion of 1g of intravenous taurine as part of the nitrogen source of parenteral nutrition reduces parenteral nutrition associated cholestatic liver disease

SECONDARY OUTCOMES:
Can additional taurine affect septic complications occuring in patients receiving parenteral nutrition
Can additional taurine improve dendritic cell function
Do patients on home parenteral nutrition have low levels of taurine
Does giving additional taurine cause an increase in levels of taurine
Does giving additional taurine cause an increase in urinary taurine excretion

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gabe, MD, Principal Investigator — North West London NHS Trust - St Mark's Hospital
Locations (1):
- North West London NHS Trust - St Mark's Hospital, Harrow, London, Middlesex, United Kingdom